CLINICAL TRIAL: NCT06634927
Title: A Randomized, Open-label, Single-dose, Parallel-controlled Phase I Clinical Trial Comparing the Pharmacokinetic Similarity, Safety, and Immunogenicity of Semaglutide Injection and Ozempic ® Injection in Healthy Subjects.
Brief Title: Pharmacokinetic Similarity, Safety, and Immunogenicity of Semaglutide Injection and Ozempic ® Injection in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HDG1901-103
Record Dates: First submitted 2024-09-24; First posted 2024-10-10 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes
Keywords: Glucagon-Like Peptide-1 Receptor Agonists; semaglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Experimental group: Semaglutide injection, specifications: 1.34 mg/mL, 1.5 mL (pre-filled injection pen), 0.25 mg , subcutaneous abdominal injection.
  Interventions: Drug: HDG1901
- Active Comparator (Active Comparator): Control group: Ozempic ® injection, 1.34 mg/mL, 1.5 mL (pre-filled injection pen), 0.25 mg , subcutaneous injection into the abdomen.
  Interventions: Drug: Ozempic®

INTERVENTIONS:
Drug: Ozempic® — Participants will be given Ozempic ® injection 0.25mg abdominal subcutaneous injection.
  Arms: Active Comparator
Drug: HDG1901 — Participants will be given HDG1901 injection 0.25mg abdominal subcutaneous injection.
  Arms: Experimental group

SUMMARY:
This study is a randomized, open-label, single-dose, parallel-controlled biosimilar comparison study comparing the pharmacokinetics, safety and immunogenicity of the investigational drug and the active comparator in healthy adult subjects. Eligible healthy participants will be screened and randomly assigned to the experimental group and the active comparator group at a ratio of 1:1 , semaglutide injection or Ozempic® injection 0.25mg abdominal subcutaneous injection will be given according to their groups. Follow-up for 5 weeks after administrtion.

Studies included a screening period (up to 2 weeks), baseline, administration (single dose), and a follow-up period (5 weeks). The duration of the study will be approximately 7 weeks for a participant.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be enrolled in the study:

1. Voluntarily participate in the trial and sign the informed consent; Willing and able, in the investigator's judgment, to comply with all experimental requirements and restrictions;
2. Healthy men and women, aged 18 to 55 years old (including);
3. Body mass index (BMI) 19.0~25.0 kg/m2 (including), weight ≥50.0 kg;
4. Physical examination, vital signs, 12-lead electrocardiogram (ECG), clinical laboratory examination, no clinically significant abnormalities;

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded:

1. Have a history of clinically serious disease or currently have any clinically significant cardiovascular, metabolic, endocrine, kidney, liver, gastrointestinal, hematological, respiratory, cutaneous, neurological, gynecological, psychiatric or other disease;
2. A history of medullary thyroid carcinoma (MTC), multiple endocrine adenoma (MEN) 2A or 2B syndrome, or related family history; Or other malignant tumor history;
3. Subjects with a history of acute and chronic pancreatitis, symptomatic gallbladder history, pancreatic injury history and other high-risk factors that may lead to pancreatitis;
4. In the screening period, calcitonin was greater than the upper limit of normal;
5. Patients with HbA1c greater than 6.5% during the screening period;
6. Those who smoked more than 5 cigarettes per day in the 3 months before screening and those who could not smoke during the whole test period;
7. Those who have a history of alcohol abuse in the six months prior to screening, or who cannot abstain from alcohol during the test period;
8. Consume any food or drink containing caffeine, alcohol, xanthine or grapefruit (such as coffee, strong tea, chocolate, etc.) within 48 hours before check-in;
9. Known or suspected allergy to semaglutide injection or similar products and excipients;
10. Participants in clinical trials of any approved or unapproved investigational drug/device within 90 days prior to screening;
11. Pregnant and lactating female subjects;
12. Patients with difficulty in venous blood collection;
13. Those who were vaccinated within 4 weeks prior to screening or planned to be vaccinated during the trial;
14. People who donate blood or lose more than 400 mL of blood or receive blood transfusions or use blood products in the 3 months prior to screening;
15. Patients who have previously received Semaglutide injection or other GLP-1 or GLP-1/ GIP-like treatment;
16. Those who have a history of drug abuse or test positive for drug abuse screening;
17. Those who test positive for blood alcohol;
18. For any other reason, the investigator does not consider the volunteer to be suitable for participation in this clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2024-09-22 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
AUC0-inf | -60minutes and 6, 12, 18, 24, 30, 36, 42, 48, 60, 72, 84, 96, 108, 120, 144, 336, 504, 672, 840 hours after administration
  Area Under the Concentration-time curve from time zero to infinite time
AUC0-t | -60minutes and 6, 12, 18, 24, 30, 36, 42, 48, 60, 72, 84, 96, 108, 120, 144, 336, 504, 672, 840 hours after administration
  Area Under the Concentration-time curve from time zero to the last measurable concentration
Cmax | -60minutes and 6, 12, 18, 24, 30, 36, 42, 48, 60, 72, 84, 96, 108, 120, 144, 336, 504, 672, 840 hours after administration
  Maximum concentration of the active substance in the blood plasma of participants during the observation period

SECONDARY OUTCOMES:
AUC_%Extrap | -60minutes and 6, 12, 18, 24, 30, 36, 42, 48, 60, 72, 84, 96, 108, 120, 144, 336, 504, 672, 840 hours after administration
  Extrapolated Part Percentage of AUC0-inf
Tmax | -60minutes and 6, 12, 18, 24, 30, 36, 42, 48, 60, 72, 84, 96, 108, 120, 144, 336, 504, 672, 840 hours after administration
  Time of maximum concentration observed
t 1/2 | -60minutes and 6, 12, 18, 24, 30, 36, 42, 48, 60, 72, 84, 96, 108, 120, 144, 336, 504, 672, 840 hours after administration
  Elimination half life
λz | -60minutes and 6, 12, 18, 24, 30, 36, 42, 48, 60, 72, 84, 96, 108, 120, 144, 336, 504, 672, 840 hours after administration
  The Volume of Distribution at Terminal Phase
CL | -60minutes and 6, 12, 18, 24, 30, 36, 42, 48, 60, 72, 84, 96, 108, 120, 144, 336, 504, 672, 840 hours after administration
  Clearance Rate
Safety and Immunogenicity | AEs will be collected after assigning the ICF. Immunogenicity sample will be collected at -60 minutes and 336、840 hours after administration.
  Adverse events and positive rate of anti-drug antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, Anhui, China